CLINICAL TRIAL: NCT05674474
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a 20-mg Dose of Vorasidenib in Subjects With Moderate or Mild Hepatic Impairment and Matched Subjects With Normal Hepatic Function
Brief Title: A Study of Vorasidenib in Participants With Moderate or Mild Hepatic Impairment and Matched Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKH-95032-008
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Impairment
Keywords: Vorasidenib
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single oral dose of 20 mg (2 × 10 mg) vorasidenib tablets on Day 1.
  Interventions: Drug: Vorasidenib
- Group B: Moderate or Mild Hepatic Impairment (Experimental): Stage 1: Participants with moderate hepatic impairment (Child-Pugh [C-P] Class B, score of 7 to 9) will receive a single oral dose of 20 mg (2 × 10 mg) vorasidenib tablets on Day 1.
  Stage 2: Participants with mild hepatic impairment (C-P Class A, score of 5 to 6) will receive a single oral dose of 20 mg (2 × 10 mg) vorasidenib tablets on Day 1. Stage 2 will be conducted if a clinically meaningful increase in exposure of vorasidenib is observed in participants with moderate hepatic impairment in Stage 1.
  Interventions: Drug: Vorasidenib

INTERVENTIONS:
Drug: Vorasidenib — Administered orally as tablets.
  Other Names: S095032; AG-881

SUMMARY:
The primary purpose of this study is to estimate the effect of moderate or mild hepatic impairment on the pharmacokinetic (PK) profile of a single oral dose of 20 mg vorasidenib in participants with hepatic impairment relative to healthy matched control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Have a body mass index of 18 to 40 kilograms per square meter (kg/m^2).
* Female participants of childbearing potential must use 2 effective methods of birth control during the study and for 90 days after the last dose of vorasidenib or be surgically sterile, or postmenopausal.
* Male participants with female partners of childbearing potential must be sterile, or willing to use 2 effective methods of birth control from Screening until at least 90 days after the last dose of the study drug, or practice abstinence during the study.
* Non-smoker or uses ≤10 cigarettes per day as judged by the investigator.
* Agree to comply with all protocol requirements for the duration of the study.
* Able to provide written informed consent prior to any procedure required by the study.

Inclusion Criteria for Healthy Participants Only:

* Have normal hepatic function.

Inclusion Criteria for Participants with Hepatic Impairment Only:

* Have chronic (more than 6 months) and stable hepatic impairment (i.e., no acute episodes of illness within 30 days before Screening due to deterioration of hepatic function) as assessed by a Child-Pugh classification score of moderate (7 to 9 points) and, if Stage 2 enrolls, mild (5 to 6 points).
* The subject has grade 0 or grade 1 hepatic encephalopathy, considered stable per investigator assessment, without exacerbation within the 6 months prior to Screening.
* The subject has a QTcF of ≤480 msec.

Exclusion Criteria for All Participants:

* Have a history or clinical manifestations of a significant neurological, renal, cardiovascular, gastrointestinal, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
* Have a history (within 5 years) or presence of malignancy, except for adequately treated basal cell and squamous cell carcinoma of the skin.
* The subject is a woman of childbearing potential who is pregnant, lactating, or planning to become pregnant within 90 days after the last dose of study drug or the subject is on oral contraceptive pills within 14 days or 5 half-lives (whichever is longer) prior to the first dose administration and during the study.
* Have received any vaccine or used any prescription (excluding hormone replacement therapy) or over-the-counter medications, including herbal or nutritional supplements, within 30 days before the first dose of the study drug.
* Have a positive test result for hepatitis B surface antigen or antibodies to hepatitis C virus.
* Have a positive test result for the presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Have a positive test result for human immunodeficiency virus (HIV) types 1 or 2 antibodies.
* Have used strong or moderate CYP1A2 inhibitors and/or inducers within 14 days or 5 half-lives, whichever is longer, prior to the first dose administration. .
* Have used any gastric acid reducing agents (eg, proton-pump inhibitors, H2-receptor antagonists, antacids) or drugs that can prolong the QT interval for 28 days or 5 drug half-lives (whichever is longer) prior to the first dosing and throughout the study
* Have a history of severe and/or uncontrolled ventricular arrhythmias or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome).
* Have a history of alcoholism or drug abuse within 3 months before Screening or excessive alcohol consumption.
* Unable or unwilling to abstain from recreational drugs, alcohol, caffeine, xanthine-containing beverages or food (e.g., coffee, tea, chocolate, and caffeinated sodas, colas), grapefruit, grapefruit juice, Seville oranges, or products containing any of these, from 48 hours prior to study drug dosing until discharge.
* Involved in strenuous activity (i.e., >30 minutes [min] per day) or contact sports within 48 hours of the first dose of the study drug or during the study.
* Have a history of relevant drug and/or food allergies (i.e., allergy to drugs with the same class effect as vorasidenib or any excipients, or any significant food allergy).
* Have received study drug in another investigational study within 30 days of dosing.

Exclusion Criteria for Participants with Hepatic Impairment Only:

* Have ascites that requires paracentesis every 4 weeks or less frequently.
* Have evidence of hepatorenal syndrome or hepatic encephalopathy.
* Have a history of incipient/planned liver transplantation within 6 months of Screening or have received a liver transplant.
* Have amylase and/or lipase levels ≥3 x upper limit of normal (ULN). Presence of 8 x ULN elevations in aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin and international normalized ratio (INR) of 3.5 for the hepatic impaired group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-t) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
AUC From Time 0 Extrapolated to Infinity (AUC0-inf) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose

SECONDARY OUTCOMES:
Apparent Terminal Elimination Half-life (t1/2) of Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Apparent Oral Clearance (CL/F) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Apparent Volume of Distribution (Vz/F) of Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Area Under the Unbound Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-t,u) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Area Under the Unbound Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUCinf,u) for Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Maximum Observed Unbound Plasma Concentration (Cmax,u) of Vorasidenib | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Cmax of Metabolite AGI-69460 | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Tmax of Metabolite AGI-69460 | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
AUC0-t for Metabolite AGI-69460 | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
AUC0-inf for Metabolite AGI-69460 | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
Number of Participants With Adverse Events (AEs) | Up to end of study [EOS] (up to approximately 29 days)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered an investigational medicinal product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Number of Participants With Abnormalities in Laboratory Parameters | Up to EOS (up to approximately 29 days)
  Clinical laboratory assessments will include hematology, serum chemistry, coagulation, and urinalysis.
Number of Participants With Abnormalities in Vital Signs | Up to EOS (up to approximately 29 days)
  Systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature will be assessed.
Number of Participants With Abnormalities in 12-Lead Electrocardiogram (ECG) Results | Up to EOS (up to approximately 29 days)
Number of Participants With Abnormalities in Physical Examination Findings | Up to EOS (up to approximately 29 days)

CONTACTS AND LOCATIONS:
Locations (1):
- American Research Corporation, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  sponsored by Servier with a first patient enrolled as of 1 January 2004 onwards for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/